CLINICAL TRIAL: NCT03544567
Title: A Phase 2 Study of Oraxol in Subjects With Cutaneous Angiosarcoma
Brief Title: A Study of Oraxol in Subjects With Cutaneous Angiosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KX-ORAX-010
Record Dates: First submitted 2018-04-05; First posted 2018-06-04 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-01

CONDITIONS: Angiosarcoma of Skin
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oraxol (Experimental): Oraxol will be administered once daily for 3 consecutive days every week from Weeks 1 through 25. Subjects who do not have documented disease progression by the end of the Treatment Period will be eligible to receive therapy in the Treatment Extension Period; additional doses of Oraxol may be administered from Week 26 onwards. Subjects may receive Oraxol until they meet 1 of the criteria for withdrawal from the study.
  Interventions: Drug: Oraxol

INTERVENTIONS:
Drug: Oraxol — oral paclitaxel will be supplied in capsules and oral HM30181A-US in tablets
  Other Names: oral HM30181A + oral paclitaxel

SUMMARY:
This is a non-blinded, multi-center, open-label, phase 2 study to evaluate the activity, safety, and tolerability of Oraxol in subjects with cutaneous angiosarcoma.

DETAILED DESCRIPTION:
Oraxol will be administered once daily for 3 consecutive days every week during the Treatment Period from Weeks 1 through 25.

Subjects who do not have documented disease progression by the end of the Treatment Period will be eligible to receive therapy in the Treatment Extension Period; Oraxol may be administered from Week 26 onwards.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to give informed consent, prior to any study-specific procedures and willingness to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
* Age of 18 years or older
* Histologically-confirmed cutaneous angiosarcoma that is not amenable to curative intent surgery (eg, locally advanced disease and disease for which surgical resection would carry an unacceptable risk of recurrence or morbidity to the subject)
* Subjects who have not received taxanes for the treatment of angiosarcoma
* Measurable disease per RECIST v.1.1
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Resolution of all acute AEs resulting from prior cancer therapies to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 (NCI CTCAE v4.03) Grade ≤1 or to that subject's baseline
* Adequate organ function as defined by the following criteria:

  * Adequate renal function as evidenced by serum creatinine ≤1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥50 mL/min per the Cockcroft and Gault formula
  * Adequate bone marrow function as evidenced by:

    * absolute neutrophil count (ANC) ≥1.5 × 109/L
    * hemoglobin ≥9.0 g/dL (<9.0 g/dL is acceptable if it is corrected by transfusion), and
    * platelet count ≥100 × 109/L
  * Adequate liver function as evidenced by

    * total bilirubin within normal limits,
    * alanine aminotransferase (ALT) ≤3×ULN, and aspartate aminotransferase (AST) ≤3×ULN,
    * gamma-glutamyl transferase (GGT) ≤10×ULN, and
    * alkaline phosphatase ≤3×ULN
* Able to swallow pills whole and retain oral medications
* Sexually active male subjects including men who are sterile (including vasectomy confirmed by post vasectomy semen analysis) must agree to use a condom with spermicide and to not donate sperm from the time of Screening until 6 months following the last dose of Oraxol
* Women of non-child bearing potential due to surgical sterilization (at least 6 weeks following surgical bilateral oophorectomy with or without hysterectomy or tubal ligation) confirmed by medical history or menopause (ie, no menstrual bleeding for more than 12 months in a woman aged ≥45 years), OR women of childbearing potential who test negative for pregnancy at time of enrollment based on serum pregnancy test must be using a highly effective method of contraception from the time of Screening until 6 months following the last dose of Oraxol. Note: Highly effective methods of contraception that result in a low failure rate (ie, <1% per year) when used consistently and correctly include combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner, or sexual abstinence. True abstinence, when in line with the preferred and usual lifestyle of the subject, is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of study participation and for 6 months post-Oraxol administration. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the subject. Periodic abstinence (eg, calendar, ovulation, symptothermal, and post-ovulation method) and withdrawal are not acceptable methods of contraception.
* Life expectancy of at least 3 months, in the opinion of the Investigator

Exclusion Criteria:

* Subjects with metastases outside of local lymph node involvement
* Concurrent treatment or participation on other therapeutic clinical trial for angiosarcoma. Participation in companion studies sponsored by local institutions, including biological correlates, is permitted.
* Women who are pregnant or breastfeeding
* Receipt of systemic cytotoxic therapy, including investigational agents, within 14 days or 5 half-lives of the first study dosing day, whichever is longer
* Major surgery or trauma within 28 days prior to first dose of investigational product. Note: The following are not considered to be major procedures and are permitted before treatment administration: thoracentesis, paracentesis, catheter placement, port placement, laparoscopy, thoracoscopy, tube thoracostomy, bronchoscopy, endoscopic ultrasonographic procedures, mediastinoscopy, skin biopsies, and imaging-guided biopsy for diagnostic purposes
* Subjects who have received wide-field radiotherapy to the pelvis ≤3 months (defined as >50% of volume of pelvic bones or equivalent) or limited-field radiation for palliation ≤3 months prior to treatment administration. Angiosarcoma lesions in the radiation field are not evaluable unless they have developed progressive disease following radiation.
* History of brain involvement with cancer, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease.
* Angina, myocardial infarction, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism, pulmonary embolism, percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG) within 3 months prior to treatment administration
* Active bleeding or bleeding diathesis actively requiring transfusions; Note: subjects with cutaneous ulcers from angiosarcoma or who have skin lesions with bleeding are allowed to participate.
* Thrombolytic use (except to maintain IV catheters) within 10 days prior to treatment administration
* Presence of a malabsorption syndrome or major resection of the stomach or small bowel that could affect the absorption of Oraxol
* Known active viral or nonviral hepatitis or cirrhosis
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
* Active infection that requires systemic treatment
* Concurrent use of a strong cytochrome P450 (CYP) 3A4 inducer (eg, rifampin or St. John's Wort) or a strong CYP3A4 inhibitor (eg, ketoconazole) within 14 days prior to treatment administration
* Concurrent use of a strong CYP2C8 inhibitor (eg, gemfibrozil) or inducer (eg, rifampin) within 14 days prior to treatment administration
* Concurrent use of an oral medication with a narrow therapeutic index known to be a P-glycoprotein (P-gp) substrate within 24 hours prior to treatment administration
* Concurrent use of a medication known to be a strong P-gp inhibitor or inducer within 14 days prior to treatment administration
* History of hypersensitivity to paclitaxel, not attributed to a hypersensitivity-type reaction to Cremophor® or history of hypersensitivity-type reaction to polysorbate 80 or other components of the formulation of Oraxol
* Other severe acute or chronic medical (including bone marrow suppressive diseases) or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation, impede the ability of the subject to complete all protocol-specified activities, or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for this study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 months
  To determine the response rate 6 months after initiation of treatment with Oraxol in subjects with cutaneous angiosarcoma

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | an average of 1 year
  Overall safety and tolerability of Oraxol in subjects with cutaneous angiosarcoma
Progression free survival | 36 months
  To determine the progression-free survival (PFS) after initiation of treatment with Oraxol in subjects with cutaneous angiosarcoma
Overall Survival (OS) | 36 months
  To determine the overall survival (OS) after initiation of treatment with Oraxol in subjects with cutaneous angiosarcoma
Duration of response | 36 months
  To determine the duration of response in subjects with cutaneous angiosarcoma
Time to best response | an average of 1 year
  To determine the time to best response in subjects with cutaneous angiosarcoma
Progression Free Rate | 6 months
  To determine the progression free rate at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Cutler, MD, Study Director — Athenex, Inc.
Locations (10):
- United States (4):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Texas Oncology, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Washington/Fred Hutchinson Cancer Center, Seattle, Washington
- Prince of Wales Hospital, Shatin, Hong Kong, Hong Kong
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hosptial, Taipei
- United Kingdom (3):
  - University College London Hospitals NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester, Manchester

IPD SHARING:
Plan to Share IPD: No